CLINICAL TRIAL: NCT05203900
Title: An Investigation of the Influence by Dietary Human Milk Oligosaccharide on Growth Factors and Cytokines in Blood, and Gut Microbiota in Low Birth Weight Infants (a Non-blinded Pilot Clinical Study)
Brief Title: The Influence by Dietary Human Milk Oligosaccharide in Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meiji Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-003
Record Dates: First submitted 2021-12-23; First posted 2022-01-24 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-02

CONDITIONS: Low Birth Weight Infants
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: The number of anticipated participants is 60 mother-infant pairs. The 30 first enrolled mother-infant pairs are assigned to the investigational formula group, and the next 30 enrolled mother-infant pairs are assigned to the control formula group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational formula (Experimental): Infant formula with Human Milk Oligosaccharide
  Interventions: Dietary Supplement: Infant formula with Human Milk Oligosaccharide
- Control formula (Placebo Comparator): Infant formula without Human Milk Oligosaccharide
  Interventions: Dietary Supplement: Infant formula without Human Milk Oligosaccharide

INTERVENTIONS:
Dietary Supplement: Infant formula with Human Milk Oligosaccharide — Although breastfeeding is encouraged, the shortage is supplemented with the investigational formula. After obtaining the informed consent, the investigational formula is administered to infants under the doctor's direction until a medical check-up at one-month-old.
  Arms: Investigational formula
Dietary Supplement: Infant formula without Human Milk Oligosaccharide — Although breastfeeding is encouraged, the shortage is supplemented with the control formula. After obtaining the informed consent, the control formula is administered to infants under the doctor's direction until a medical check-up at one-month-old.
  Arms: Control formula

SUMMARY:
This study aims to investigate the concentration of various growth factors and cytokines in blood, and to examine the gut microbiota of low birth weight infants fed with formulas with or without Human Milk Oligosaccharide (HMO) supplement. Eligible low birth weight infants are allocated to two groups, Investigational formula (with HMO) or Control formula (without HMO). The subjects are taking the assigned formula when they need to be supplemented with formula. After the informed consent was obtained and eligibility was confirmed, the intervention period begins, and ends at the one-month-old medical check-up with the assessment of the various blood growth factors and cytokines, and the gut microbiota.

ELIGIBILITY:
1. Inclusion Criteria:

   1-1) For infants

   i. Low birth weight infants (defined as a birth weight ≥1,500 g and <2,500 g) during hospitalization and may require milk powder formula as supplement.

   1-2) For mothers

   i. Mothers who do not find serious viral infection

   ii. Mothers who are willing to provide consent for provision of study required information and specimen(s) from both mothers and infants

   iii. Mothers who are willing to provide consent as infant's legally acceptable representative (LAR)
2. Exclusion Criteria:

   2-1) For infants

   i. Infants who receive any formulas before Informed Consent.

   ii. Infants with serious infections.

   iii. Infants with necrotizing enteritis.

   iv. Infants with gastrointestinal perforation.

   v. Infants whom the PI determines inappropriate as a study subject (e.g. inflammatory, metabolic abnormalities and difficulty in enteral feeding).

   2-2) For mothers

   i. Mothers the PI determines inappropriate as a study subject

   ii. Mothers under 18 years old.
3. Withdrawal criteria:

A subject must be discontinued from treatment with test formula if any of the following apply:

i. If the mother, who is a subject of the study as well as infant's LAR , asks for withdrawal from the study or withdraws consent.

ii. When a serious adverse event occurs.

iii. When an adverse event occurs, and the PI or co-investigator determines that the study should be discontinued.

iv. If it is decided that there is a risk of compromising the safety of the study subject.

v. If a subject is found to be ineligible after the start of the study.

vi. If it is found that there is a serious or continued non-compliance with the study protocol by a study subject.

vii. In addition, if the PI decides to end the study.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Growth factors concentration in infant's plasma | At one-month-old
  The concentration of NGF-beta (pg/mL), BDNF (pg/mL), etc. in infant's plasma will be measured by immunoassay.
Cytokines concentration in infant's plasma | At one-month-old
  The concentration of IFN-gamma (pg/mL), IL-1alpha (pg/mL), etc. in infant's plasma will be measured by immunoassay.
Infant's gut microbiota occupancy | At one-month-old
  Total bacterial counts and bifidobacterial counts in stool will be measured by RT-PCR (copy/g wet feces). Occupancy of microbiota in infant's stool will be comprehensively analyzed by DNA/RNA Sequencing (percent).

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No